CLINICAL TRIAL: NCT07273994
Title: Multicenter Randomized Clinical Trial To Evaluate Two Different Amiodarone Regimens To Maintain Sinus Rhythm After Electrical Cardioversion In Persistent Atrial Fibrillation
Brief Title: Evaluation of Two Different Regimens of the Antiarrhythmic Drug Amiodarone to Maintain Normal Sinus Rhythm After Electrical Cardioversion in Patients With Persistent Atrial Fibrillation
Acronym: PERIVERSION-2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-AMI-2024-33; Project PI023/1768 (Other Grant/Funding Number: Instituto Salud Carlos III, Ministry of Science, Innovation and Universities, Government of Spain.); 2024-514113-35-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-19; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-03

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Atrial fibrillation; Electrical cardioversion; Amiodarone; Pharmacogenetics; Adverse effects
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amiodarone full doses (Active Comparator): Patients will receive amiodarone full doses (200 mg/day) (Usual dose)
  Interventions: Drug: Amiodarone Hydrochloride 200 MG
- Amiodarone reduced doses (Experimental): Patients will receive amiodarone reduced doses (100 mg/day)
  Interventions: Drug: Amiodarone Hydrochloride 100 MG

INTERVENTIONS:
Drug: Amiodarone Hydrochloride 200 MG — Patients will receive full amiodarone daily doses: 200 mg/day
  Arms: Amiodarone full doses
Drug: Amiodarone Hydrochloride 100 MG — Patients will receive amiodarone reduced daily doses: 100 mg/d
  Arms: Amiodarone reduced doses

SUMMARY:
---

The goal of this clinical trial is to learn if reduced doses of amiodarone can treat atrial fibrillation (AF) effectively while minimizing toxic side effects in patients with persistent AF after electrical cardioversion. The main questions it aims to answer are:

* Can a reduced dose of amiodarone (100 mg/day) maintain sinus rhythm as effectively as the standard dose (200 mg/day) 12 months post electrical cardioversion?
* What are the adverse effects of the standard and reduced doses of amiodarone during 12 months post electrical cardioversion?
* How do genetic polymorphisms affect the efficacy and safety of amiodarone?
* How do amiodarone plasma levels correlate with the maintenance of sinus rhythm and genetic polymorphisms?

Researchers will compare the standard dose (200 mg/day) to the reduced dose (100 mg/day) to see if the reduced dose offers a better balance between efficacy and safety.

Participants will:

* Be treated with full dose amiodarone (200 mg/day) during the first month after electrical cardioversion.
* Be randomized to either continue with the full dose (200 mg/day) or switch to the reduced dose (100 mg/day).

The study is a multicenter, randomized clinical trial involving 312 patients with persistent AF after successful electrical cardioversion. Participants will be followed for 12-18 months to monitor the recurrence of AF and adverse effects.

ELIGIBILITY:
Inclusion Criteria

1. Patients aged ≥ 18 years
2. Documented persistent atrial fibrillation (≥ 7 days in duration)
3. Electively referred for Electrical Cardioversion
4. Signed informed consent.

Exclusion Criteria

1. Urgent electrical cardioversion
2. Atrial fibrillation post-cardiac surgery
3. Previous myocardial infarction
4. New York Heart Association (NYHA) Class IV heart failure
5. Left ventricular ejection fraction (LVEF) <45%
6. Significant left ventricular hypertrophy (wall thickness ≥ 15mm)
7. Hyperthyroidism or hypothyroidism
8. Known hepatobiliary disease (acute hepatitis, cirrhosis...) or ALT/AST > 3 x upper limit of normal (ULN)
9. Allergy, intolerance, or known hypersensitivity to study medications
10. Women of childbearing potential unwilling to use contraceptive measures and breastfeeding women.
11. Participation in another clinical trial involving investigational drugs
12. Life expectancy less than 12 months
13. Rheumatic mitral stenosis of any degree or severe mitral or aortic valve dysfunction.
14. Patients with contraindications to amiodarone, such as uncontrolled thyroid dysfunction, severe sinus bradycardia, second- or third-degree AV block without a pacemaker, and a history of amiodarone-induced pulmonary toxicity.
15. Patients in whom chronic amiodarone treatment previously failed to maintain sinus rhythm
16. Patients with abnormal baseline QTc (>450 ms in males and >470 in females) or abnormal ECG that precludes QTc assessment
17. Patients requiring concomitant medications that have a higher risk of QTc prolongation.
18. Patient do not have a smart mobile phone or do not know how to use it adequately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Maintenance of sinus rhythm | 12 months follow-up
  Number of patients mantaining sinus rhythm 12 months post electrical cardioversion

SECONDARY OUTCOMES:
Adverse effects | 12 months follow-up
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Polymorphisms | 12 months follow-up
  Association of the different assessed polymorphisms with the primary and first secondary outcome
Plasma levels | 12 months follow-up
  Correlation of amiodarone plasma levels during follow-up with the maintenance of sinus rhythm

OTHER OUTCOMES:
Plasma levels - polymorphisms | 12 month follow-up
  Correlation of amiodarone plasma levels with polymorphisms

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No